CLINICAL TRIAL: NCT01875302
Title: Comparison of an Electronic Version of Selected COPD PRO Instruments With the Original Versions
Status: Completed | Type: Observational
Sponsor: nSpire Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NSH-001
Record Dates: First submitted 2013-04-22; First posted 2013-06-11 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: COPD
Keywords: COPD PRO Instraments equivalency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol defines the requirements to demonstrate that the PRO instruments which were designed as paper-based are equivalent to the nSpire Health ePRO (electronic patient reported outcome), following the ISPOR's ePRO Good Research Practices Task Force recommendations. All validation studies of the questionnaires were conducted using the original paper versions.

ELIGIBILITY:
Inclusion Criteria:

* Give their signed written informed consent to participate
* Current symptoms COPD, as diagnosed by a physician
* Age 40 - 75 years
* Able to read and understand English

Exclusion Criteria:

• Unwilling to complete the 3 electronic PRO questionnaires or participate in an interview during completion of questionnaires

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD Subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Demonstrate that the following PRO instruments which were designed as paper-based are equivalent to the nSpire Health ePRO (electronic patient reported outcome) | 60 minutes
  The primary measures to demonstrate equivalency of electronic to paper PRO instruments are Usability and Cognitive Debriefing.
  Usability data is gathered using systematic observation under controlled conditions to determine how well the device may be used by subjects.
  Qualitative, Content Analysis of Cognitive Debriefing Data The cognitive debriefing data will be content analyzed for subject understanding of the instructions on the device used to deliver the PRO instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Vig, MS, Study Director — nSpire Health